CLINICAL TRIAL: NCT05269004
Title: A Multicenter, Single-Arm, Open-Label, Extension, Rollover Study To Evaluate The Long-Term Safety And Efficacy Of Ocrelizumab In Patients With Multiple Sclerosis
Brief Title: A Rollover Study to Evaluate the Long-Term Safety and Efficacy of Ocrelizumab In Patients With Multiple Sclerosis
Acronym: OLERO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MN43964; 2021-005746-15 (EudraCT Number)
Record Dates: First submitted 2022-02-11; First posted 2022-03-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab (Experimental): Participants receiving ocrelizumab as an investigational medicinal product (IMP) in a Roche sponsored Parent study who continue to receive ocrelizumab or are in safety follow-up at the time of the closure of their respective Parent study (WA21092, WA21093 or WA25046). Participants who will continue ocrelizumab treatment will receive IMP based on the dosage and administration received at the time of rollover from the Parent study.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered based on the dosage and administration received at the time of rollover from the Parent study.

SUMMARY:
This is a Phase IIIb, single-arm, multicenter, OLE study. Participants receiving ocrelizumab as an investigational medicinal product (IMP) in a Roche sponsored Parent study who continue to receive ocrelizumab or are in safety follow-up at the time of the closure of their respective Parent study (WA21092, WA21093 or WA25046) are eligible for enrollment in this extension study. Participants who will continue ocrelizumab treatment will receive IMP based on the dosage and administration received at the time of rollover from the Parent study.

ELIGIBILITY:
Inclusion criteria

* Prior eligibility for and previous participation in 1 of the Roche-sponsored Parent Studies WA21092, WA21093, or WA25046 with the participant either receiving ocrelizumab as an investigational medicinal product (IMP) or being in safety follow-up after treatment discontinuation
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate acceptable contraception during the treatment period and for at least 6 months or longer if the local label is more stringent after the final dose of ocrelizumab, as applicable in the ocrelizumab package leaflet

Exclusion criteria

* Concurrent participation in any clinical trial (other than the Parent study)
* Unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events, with severity determined according to the NCI CTCAE v5.0 | Up to 44 months

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score over time | Week 0, 24, 48, 72, 96, 120, 168
Change in 9-Hole Peg Test (9HPT) over time | Week 0, 24, 48, 72, 96, 120, 168
Change in Timed 25-Foot Walk Test (T25FWT) over time | Week 0, 24, 48, 72, 96, 120, 168
The number of T1 lesions and number of new or enlarging T2 lesions | Week 0, 24, 48, 72, 96, 120, 168
The change in total volume of T2 lesions and in total non-enhancing T1 lesion volume | Week 0, 24, 48, 72, 96, 120, 168

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (233):
- United States (49):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arizona Neuroscience Research LLC, Phoenix, Arizona
  - MS Center of California, Laguna Hills, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado - Anschutz Medical Campus (University of Colorado Health Sciences Center), Aurora, Colorado
  - Advanced Neurosciences Research LLC, Fort Collins, Colorado
  - Neurology Associates PA, Maitland, Florida
  - University of Miami, Miami, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Vero Beach Neurology and Research Institute, Vero Beach, Florida
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - Indiana Univ School of Med, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers New Jersey Medical School Department of Neurology, Newark, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - South Shore Neurologic Associates PC, Patchogue, New York
  - SUNY at Stony Brook, Stony Brook, New York
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - The Neurological Institute PA, Charlotte, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - University Neurology Inc., Cincinnati, Ohio
  - Columbus Neuroscience, Westerville, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Providence Neurological Specialties, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Neurology Clinic PC, Cordova, Tennessee
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Uni of Texas Health Science Center At Houston, Houston, Texas
  - Bhupesh Dihenia M.D. P.A., Lubbock, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Swedish Neuroscience Institute, Seattle, Washington
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
- Argentina (2):
  - Hospital Español, Ciudad Autonoma Bs As
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Barmherzige Brueder Konventspital, Linz
  - AKH - Medizinische Universität Wien, Vienna
- Belarus (3):
  - Grodno University Hospital, Grodno, Brest Oblast
  - State Institution Minsk Research and Practice Center of Surgery Transplantation and Hematology, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Belgium (5):
  - AZ Sint Jan, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - Algemeen Ziekenhuis Alma, Eeklo
  - AZ Delta Campus Westlaan, Roeselare
- Brazil (6):
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goinia, Goiás
  - Hospital So Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - IMV Pesquisa Neurologica Sociedade Simples Ltda, Porto Alegre, Rio Grande do Sul
  - Clinica Neurológica e Neurocirúrgica de Joinville, Joinville, Santa Catarina
  - Hospital Universitario Gaffree e Guinle, Rio de Janeiro
  - HUCFF-UFRJ - Hospital Universitário Clementino Fraga Filho Universidade Federal do Rio de Janeiro, Rio de Janeiro
- Bulgaria (6):
  - MHAT Avis Medica OOD Department of Neurology, Pleven
  - MHATNP Sveti Naum EAD, Sofia
  - University First MHAT-Sofia St. Joan Krastitel EAD, Sofia
  - National Heart Hospital EAD, Sofia
  - Acibadem City Clinic Tokuda Hospital Ead, Sofia
  - Military Medical Academy MHAT Sofia Department of Rheumatology, Sofia
- Canada (8):
  - Calgary MS Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - UBC Multiple Sclerosis & Neuromyelitis Optica NMO Clinical Trials, Vancouver, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - St Michael Hospital, Toronto, Ontario
  - Clinique Neuro Outaouais, Gatineau, Quebec
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Croatia (2):
  - General Hospital Varazdin, Varaždin
  - University Hospital Center Zagreb, Zagreb
- Czechia (8):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Neurospol s.r.o., Havirov-Podlesi
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Pardubicka krajska nemocnice a.s., Pardubice
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Krajska zdravotni a.s. - Nemocnice Teplice o.z., Teplice
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Tammer Tutka Oy, Tampere, Finland
- France (9):
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen, Calvados
  - CHU Nancy Hôpital Central, Nancy, Meurthe Et Moselle
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Neurologique Pierre Wertheimer, Bron
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Roger Salengro Service de Neurologie, Lille
  - CHU Nice - Hôpital Pasteur 2, Nice
  - Centre Hospitalier Intercommunal de Poissy, Poissy
  - CHU Strasbourg Hpital Hautepierre, Strasbourg
- Germany (17):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Bayreuth GmbH, Bayreuth, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede, Lower Saxony
  - Universitaetsklinikum Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - Pharmakologisches Studienzentrum, Chemnitz, Saxony
  - Universitaetsklinikum Leipzig, Leipzig, Saxony
  - Charité Universitaetsmedizin Berlin - Campus Ch, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - Neurologie in Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Zentrum fuer ambulante Neurologie, Essen
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Universitaetsklinikum Muenster, Münster
  - Medizinische Einrichtungen des Bezirks Oberpfalz GmbH, Regensburg
- Hungary (3):
  - S-Medicon Egeszsegugyi Szolgaltato Kft., Budapest
  - Jahn Ferenc Del-Pesti Korhaz es Rendelointezet, Budapest
  - Pecsi Tudomanyegyetem, Pécs
- Israel (4):
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Azienda Socio Sanitaria Territoriale della Valle Olona (pres, Gallarate, Aosta Valley
  - Ospedale degli Infermi, Ponderano, Friuli Venezia Giulia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea-Universitr di Roma La Sapien, Rome, Lazio
  - IRCCS AOM Azienda Ospedaliera Metropolitana, Genoa, Liguria
  - Ospedale San Raffaele, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Montichiari, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Fondazione Istituto G. Giglio di Cefalu, Cefalù, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona, The Marches
- Latvia (2):
  - Maritime Medicine Centre of Latvia Hospital of Vecmilgravis Department of Neurology, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics Public Institution, Kaunas
  - Klaipeda University Hospital Public Institution, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (8):
  - Hospital Mexico Americano, Guadalajara, Mexico CITY (federal District)
  - Mexico Centre for Clinical Research, Mexico City, Mexico CITY (federal District)
  - Clinical Research Institute, Tlalnepantla, Mexico CITY (federal District)
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro de Estudios Clinicos y Especialidades Medicas S C, Monterrey, Nuevo León
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Hospital Angeles Chihuahua, Chihuahua City
  - Grupo Medico Camino, México
- Zuyderland Medisch Centrum - Sittard-Geleen', Sittard-Geleen, Netherlands
- Waikato Hospital, Hamilton, New Zealand
- Haukeland Universitetssykehus, Bergen, Norway
- Poland (12):
  - NZOZ Vitamed, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp z o o, Gda?sk
  - M.A. LEK A.M.Maciejowscy SC., Katowice
  - Specjal. Praktyka Lekarska, Katowice
  - Neuro-Medic Janusz Zbrojkiewicz, Katowice
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - Neurologiczny NZOZ Centrum Leczenia SM, Plewiska
  - Neuro-Care Gabriela Klodowska, Siemianowice ?l?skie
  - Centrum Medyczne NeuroProtect, Warsaw
- Portugal (4):
  - Centro Clnico Acadmico - Braga, Associao (2CA-Braga), Braga
  - Centro Hospitalar do Porto, E.P.E. - Hospital de Santo Antnio, Coimbra
  - Unidade Local de Saude de Santa Maria, E.P.E. - Hospital de Santa Maria, Lisbon
  - Hospital Garcia de Orta, Pragal
- Romania (2):
  - Spitalul Universitar de Urgenta Elias, Bucharest
  - SC Clubul Sanatatii SRL, Campulung Muscel
- Russia (18):
  - Siberian Medical Center, Barnaul, Altayskiy Kray
  - FSBI 'Federal Scientific and Clinical Center of Specialized Types of Medical Care and Medical Techno, Moscow, Moscow Oblast
  - SBIH City Polyclinic 2 of the Department of Health of the City of Moscow, Moscow, Moscow Oblast
  - SBIH of Republic Mordoviya "Republican Clinical Hospital # 4", Saransk, Respublika Mordoviya
  - FSBMEI HPE "Military Medical Academy n.a. S.M. Kirov" of the MoD of the RF, Saint Petersburg, Sankt-Peterburg
  - SPb SBIH "City Multy-field Hospital # 2", Saint Petersburg, Sankt-Peterburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg, Sankt-Peterburg
  - SBIH of Stavropol territory " City Hospital # 2" of Pyatigorsk, Pyatigorsk, Stavropol Kray
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg, Sverdlovsk Oblast
  - Regional Multiple Sclerosis Centre b/o CC ECM Neftyanik, Tyumen, Tyumen Oblast
  - SAHI "Interregional Clinical and Diagnostic Center", Kazan, Vologda Oblast
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - Kirov RSBIH "Kirov City Clinical Hospital # 1", Kirov
  - FSBIH Siberian Clinical Center of FMBA of Novosibirsk, Novosibirsk
  - SBEI HPE " Perm State Medical University n.a. Academician E.A. Vagner" of the MoH of the RF, Perm
  - SBEI HPE "Samara State Medical University" of the MoH of the RF, Samara
  - Saratov State Medical University, Saratov
  - RSBIH "Smolensk Regional Clinical Hospital", Smolensk
- Serbia (2):
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Slovakia (3):
  - MUDr. Beata Dupejova Neurologicka ambulancia s.r.o, Banská Bystrica
  - Univerzitna nemocnica Bratislava Nemocnica Ruzinov, Bratislava
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Spain (11):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Santa Caterina, Salt, Girona
  - Complejo Hospitalario Universitario de Santiago (CHUS) Servicio de Neurologia, Santiago de Compostela, LA Coruna
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (2):
  - Sahlgrenska Sjukhuset, Gothenburg
  - Akademiskt Specialist Centrum, Stockholm
- Switzerland (2):
  - Universitaetsspital Basel, Basel
  - Ospedale Regionale di Lugano, Lugano
- Tunisia (2):
  - Hopital Razi, Mannouba
  - Hopital Universitaire Fattouma Bourguiba, Monastir
- Turkey (Türkiye) (3):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ondokuz Mayis Univ. Med. Fac., Samsun
  - Karadeniz Tecnical Uni. Med. Fac, Trabzon
- Ukraine (9):
  - Medical Center of Limited Liability Company Medical Center Saliutem, Vinnytsia, Chernihiv Governorate
  - Separated structural unit ?University hospital? of Dnipro State Medical University, Dnipro, Dnipropetrovsk Oblast
  - Institute of Neurology Psychiatry and Narcology of NAMS of Ukraine, Kharkiv, Kharkiv Governorate
  - Communal noncommercial enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv, Kharkiv Governorate
  - CMPI Chernihiv Regional Hospital, Chernihiv, KIEV Governorate
  - CNE Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk, KIEV Governorate
  - Medical Center of Limited Liability Company Medbud-Clinic, Kyiv, KIEV Governorate
  - CNE of Lviv Reg Clin Hospital Dept of Neurology D.Halytskyi Lviv NMU, Lviv, KIEV Governorate
  - CNE Odesa Regional Clinical Hospital of Odesa Regional Council, Odesa, KIEV Governorate
- United Kingdom (6):
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham, Nottinghamshire
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Walton Centre For Neurology and Neurosurgery, Liverpool
  - Barts Health NHS Trust, London
  - Royal Victoria Infirmary, Newcastle
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing